CLINICAL TRIAL: NCT01887379
Title: Characterisation of Gastric Residence of a Furosemide-containing New Gastric Retention System by Means of MMM Measurement and Determination of Pharmacokinetics, Pharmacodynamics and Safety
Brief Title: Magnetic Marker Monitoring of Furosemide-containing Gastroretentive Formulation in Healthy Male Subjects (Fasting and Fed Conditions)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LTS Lohmann Therapie-Systeme AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LTS 03/10; 2013-001063-23 (EudraCT Number)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Gastroretentive Drug Formulation of Furosemide; Oedema
Keywords: Gastroretentive drug formulation; Furosemide; Magnetic Marker Monitoring; Magnetic marker; Oedema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRDF furosemide fasting conditions (Experimental): Subjects will be tested under fasting conditions after administration of GRDF Furosemide.
  Interventions: Drug: GRDF furosemide
- GRDF furosemide fed conditions (Experimental): Subjects will be tested under fed conditions after administration of GRDF Furosemide.
  Interventions: Drug: GRDF furosemide

INTERVENTIONS:
Drug: GRDF furosemide — The GRDF furosemide tablet contains Fe3O4, which serves as an inactive magnetic marker to allow monitoring of the tablet transit through the gastrointestinal tract, using the MMM imaging technique.
  Other Names: GRDF furosemide is a gastro retentive dosage form of furesomide

SUMMARY:
Furosemide is a diuretic drug, used in the treatment of oedematous states associated with cardiac, renal, and hepatic disorder, and may be effective in patients unresponsive to thiazide diuretics. Furosemide is also used in the treatment of hypertension.

Absorption of furosemide from the gastrointestinal tract is fairly rapid; bioavailability is 60-70%, but variable and not predictable, with large intra- and inter-individual variability, and are influenced by dosage form, underlying diseases, and by the presence of food after oral administration. Data from animal model show that furosemide administered into the stomach is more rapidly absorbed than if is administered into the small intestine.

To increase the residency of furosemide in the stomach after oral administration, a gastroretentive dosage form (GRDF) of furosemide has been developed. In the current study, the new formulation (30mg furosemide coated tablet) will be tested in healthy male subjects. Absorption will be characterised by an effective and safe imaging technique - Magnetic Marker Monitoring (MMM), based on Fe3O4 added to the drug product to generate magnetic signal that can be used for up to 12 h after furosemide administration to localize the medication in the gastrointestinal tract. Fe3O4 is frequently used as colouring pigment in medicinal products. It does not exhibit own pharmacodynamic activity and is considered as an inactive ingredient.

In the current study, GRDF formulation of furosemide will be evaluated for: gastric residence as well as pharmacokinetic and pharmacodynamic characteristics under fasting and fed conditions. As part of the study, the subjects will be hospitalized for 1 day during each drug administration. The duration of the stay will depend on the intestinal behaviour of the investigational product.

DETAILED DESCRIPTION:
Furosemide is a diuretic drug, widely used in the treatment of oedematous states associated with cardiac, renal, and hepatic disorder, and may be effective in patients unresponsive to thiazide diuretics. Furosemide is also used in the treatment of hypertension.

Absorption of furosemide from the gastrointestinal tract is fairly rapid. Bioavailability is reported as 60-70%, but is variable and not predictable. The rate and extent of absorption show a large intra- and inter-individual variability and are influenced by dosage form, underlying diseases, and by the presence of food after oral administration. Results obtained with an animal model indicate that furosemide administered into the stomach is more rapidly absorbed than if is is administered into the small intestine.

To increase the residency of furosemide in the stomach after oral administration, a gastroretentive dosage form (GRDF) of furosemide has been developed. In this study, the new formulation(30mg furosemide coated tablet) will be tested in healthy male subjects. Absorption will be characterised by imaging technique - Magnetic Marker Monitoring (MMM), which is the most effective and safe imaging technique currently available. MMM is based on a iron-III-oxide (Fe3O4) added to the drug product to generate magnetic signal that can be used to localize the administered medication in the gastrointestinal tract.

Fe3O4 is frequently used as colouring pigment in medicinal products. It does not exhibit own pharmacodynamic activity and thus, it is considered as clinically inactive ingredient. Fe3O4 exhibits a dipole moment and thus, after magnetisation of solid oral dosage forms containing homogenously distributed Fe3O4, the product generates a magnetic signal, which can be used for localisation of the dosage form in the gastrointestinal tract by Magnetic Marker Monitoring technique.

The aim of the current study is to evaluate the GRDF formulation of furosemide for: gastric residence, pharmacokinetic and pharmacodynamic characteristics under fasting and fed conditions. As part of the study, the subjects will be hospitalized for 1 day during each drug administration (i.e. a total of two days). The duration of the stay will depend on the intestinal behaviour of the investigational product. The MMM monitoring be performed for up to 12 h after furosemide administration. For pharmacokinetic determinations, liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS) will be used to analyze furosemide in plasma.

ELIGIBILITY:
Inclusion Criteria:

1. sex: male
2. ethnic origin: Caucasian
3. age: 18 years to 55 years
4. body-mass index (BMI): > or = 19 kg/m² and < or = 27 kg/m²
5. good state of health
6. non-smoker or ex-smoker for at least 1 month
7. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety and tolerability or with gastric emptying and the gastrointestinal transport (e.g. inflammatory bowel diseases, ileus)
4. history of relevant central nervous system (CNS) and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
5. any surgery at the gastrointestinal tract, which might interfere with the safety of the test product or any stomach reduction like Bioenterics Intragastric Balloon (BIB) or gastric banding
6. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
7. known allergic reactions to sulphonamide
8. subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
9. heart rate < 50 bpm or > 90 bpm
10. systolic blood pressure of < 100 mmHg and > 140 mmHg, diastolic blood pressure of < 60 mmHg and >90 mmHg
11. laboratory values, especially for sodium, potassium, calcium, creatinine, urea, uric acid, and blood glucose out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
12. positive anti-human immunodeficiency virus-test (if positive to be verified by western blot), surface antigen of the hepatitis B virus (HBs-AG)test [if positive to be verified by test for hepatitis B Core (HBc-IgM)] or anti-hepatitis C virus-test
13. renal failure with anuria
14. coma and praecoma hepatica
15. severe hypokalemia and/or hyponatremia
16. hypovolemia or dehydration
17. subjects with manifest or latent diabetes mellitus or gout
18. subjects with cerebrovascular insufficiency or coronary heart disease
19. subjects with bladder outlet obstruction (BOO) e.g. prostatic hypertrophy, hydronephrosis or ureteral stenosis
20. hypoproteinemia
21. liver cirrhosis and simultaneous limitation of kidney function
22. acute or chronic diseases which could affect gastric emptying and the gastrointestinal transport
23. history of or current drug or alcohol dependence
24. positive alcohol or drug test at screening examination
25. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male per day
26. subjects who are on a diet which could affect gastric emptying and the gastro-intestinal transport
27. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
28. subjects with claustrophobia
29. ferromagnetic implants or any other magnetic disturbance, which can affect the Magnetic Marker Monitoring measurement
30. blood donation or other blood loss of more than 400 ml within the last two months prior to individual enrolment of the subject
31. participation in a clinical trial during the last two months prior to individual enrolment of the subject
32. regular treatment with any systemically available medication including all ototoxic medication like aminoglycosides and medication which could affect gastric emptying and the gastrointestinal transport (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists) or antibiotics
33. subjects, who report a frequent occurrence of migraine attacks
34. subjects suspected or known not to follow instructions
35. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial
36. subjects who have forfeited their own freedom by administrative or legal award, or who are under guardianship or have been admitted in a sanitary or social institution

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Residency time of GRDF furosemide in the gastrointestinal tract, evaluated with MMM technique, under fasted and fed conditions. | every 30 min for up to 12 h after drug administration; maximal observation time 12 h
  Residency time of GRDF furosemide in the gastrointestinal track will be monitored using the non-invasive MMM technique under fasted and fed conditions. Measurements will start after each administration and last until 2 hours after gastric emptying indicated by the MMM measurement, but not longer than 12 h post administration. Each observation interval for each subject will last for a minimum of 10 min followed by a break of maximum 20 min. For meal intake, a break of the MMM measuring of 30 minutes will be performed.
  Anatomical localisation within the measuring sequences will be listed for each subject and treatment
  Statistical evaluation of gastric emptying time will include: arithmetic means, medians, minimum , maximum, standard deviation.
  GRDF=Gastro retentive dosage formulation

SECONDARY OUTCOMES:
Cmax of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  Cmax = maximum concentration in plasma; GRDF=Gastro retentive dosage formulation
Cmax of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  Cmax = maximum concentration in plasma; GRDF=Gastro retentive dosage formulation
tmax of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  tmax = time to reach maximum concentration in plasma; GRDF=Gastro retentive dosage formulation
tmax of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  tmax = time to reach maximum concentration in plasma; GRDF=Gastro retentive dosage formulation
t1/2 of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  t1/2 = apparent terminal elimination half-life; GRDF=Gastro retentive dosage formulation
t1/2 of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  t1/2 = apparent terminal elimination half-life; GRDF=Gastro retentive dosage formulation
AUC0-tlast of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUC0 = area under the plasma concentration vs. time curve from dosing time to the last measurement time point with a concentration value above the lower limit of quantitation, calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations; GRDF=Gastro retentive dosage formulation
AUC0-tlast of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUC0-tlast = area under the plasma concentration vs. time curve from dosing time to the last measurement time point with a concentration value above the lower limit of quantitation, calculated by means of the linear up/log down method (linear trapezoidal rule for increases in concentration/logarithmic trapezoidal rule for decreases in concentrations; GRDF=Gastro retentive dosage formulation
AUC 0-infinity of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUC0-infinity = AUC0-tlast + AUCexpol; GRDF=Gastro retentive dosage formulation
AUC 0-infinity of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUC0-infinity = AUC0-tlast + AUCexpol; GRDF=Gastro retentive dosage formulation
AUCextrapol of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUCextrapol = AUCextrapolated = Clast/lamda; lamda = apparent terminal elimination rate constant determined by log-linear regression; GRDF=Gastro retentive dosage formulation
AUCextrapol of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacokinetic (PK) properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  AUCextrapol = AUCextrapolated = Clast/lamda; lamda = apparent terminal elimination rate constant determined by log-linear regression; GRDF=Gastro retentive dosage formulation
CL_f of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacodynamic properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  CL_f = apparent total body clearance of furosemide: dose / AUC0-∞; GRDF=Gastro retentive dosage formulation
CL_f of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacodynamic properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  CL_f = apparent total body clearance of furosemide: dose / AUC0-∞; GRDF=Gastro retentive dosage formulation
Vdz of GRDF furosemide under fasted conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacodynamic properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  Vdz = apparent volume of distribution of furosemide: dose / (AUC0-∞ x λ); GRDF=Gastro retentive dosage formulation; λ=apparent terminal elimination rate constant determined by log-linear regression
Vdz of GRDF furosemide under fed conditions | pre-dose (within 1 h prior to drug administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after drug administration.
  Characterization of the pharmacodynamic properties of GRDF furosemide, with special focus on the absorption phase of furosemide. Compare results during fasted and fed state.
  Blood samples for the determination of furosemide concentration will be taken at pre-dose (within 1 h prior to administration) and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, and 24 h after administration.
  LC-MS/MS will be used to analyze furosemide in plasma.
  Vdz = apparent volume of distribution of furosemide: dose / (AUC0-∞ x λ); GRDF=Gastro retentive dosage formulation; λ=apparent terminal elimination rate constant determined by log-linear regression
Sodium excretion over time under fasted conditions | pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
  Sodium in urine will be measured for each time interval and total sampling time. Urine will be collected and sampled during the following sample intervals: pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
Sodium excretion over time under fed conditions | pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
  Sodium in urine will be measured for each time interval and total sampling time. Urine will be collected and sampled during the following sample intervals: pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
Urine excretion over time under fasted conditions | pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
  Urine volume will be measured for each time interval and total sampling time. Urine will be collected and sampled during the following sample intervals: pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
Urine excretion over time under fed conditions | pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.
  Urine volume will be measured for each time interval and total sampling time. Urine will be collected and sampled during the following sample intervals: pre-dose (within 1 hour prior to administration), 0-2h, 2-4h, 4-8h, and 8-12h after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH, Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Berlin, Germany